CLINICAL TRIAL: NCT00286858
Title: Clinical Observations of Automatic Algorithms for Cardiac Pacing
Brief Title: Beluga - Clinical Observations of Automatic Algorithms for Cardiac Pacing
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Beluga
Record Dates: First submitted 2006-02-02; First posted 2006-02-06 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Bradycardia; Sick Sinus Syndrome; Heart Block
MeSH Terms: conditions — Bradycardia; Sick Sinus Syndrome; Heart Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Insignia Ultra and Insignia AVT — Regular AV-Delay increase to allow for intrinsic AV conduction, if present.

SUMMARY:
This study shall evaluate in daily medical practice the clinical results of the AV delay hysteresis search algorithm in patients with a INSIGNIA ULTRA or AVT pacemaker implanted for one of the three following indications: sinus node dysfunction, atrial disease (or bradycardia/tachycardia) and atrio-ventricular paroxysmal block. In addition use and outcome of automatic functions will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Dual chamber pacemaker (INSIGNIA ULTRA or AVT pacemaker), implant not older than 60 days, estimated life expectancy more than one year in case of associated illness, Age ≥ 18 years, signed patient information.

Exclusion Criteria:

* Indication for conventional treatment with ventricular resynchronisation or by implantable defibrillator during inclusion, implanted for severe permanent AVB (AVB 2/1 and complete), PR > 250 ms, implant of the device older than 60 days before the inclusion date, Heart transplant foreseen within six months, unexplained syncope.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with indication for a dual chamber pacemaker and not having a complete AV-block are invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 903 (Actual)
Dates: Start 2006-09; Primary Completion 2009-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Impact of Atrio-ventricular hysteresis algorithm on percentage of Ventricular pacing | At 12 Months
  % Vp is compared between patients with atrio-ventricular hysteresis algorithm ON and OFF in patients with sino-atrial disease or paroxysmal AV block.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier THOMAS, MD, Principal Investigator — Clinique Ambroise Paré
Locations (40):
- France (39):
  - CHRU- Hôpital Nord, Amiens
  - Clinique Cardiologique Aressy, Aressy
  - Clinique du Lac et d'Argonay, Argonay
  - CH d'Arles, Arles
  - Clinique Paulmy, Bayonne
  - CH Beauvais, Beauvais
  - Polyclinique Bordeaux-Cauderan, Bordeaux
  - Clinique des Cèdres, Brive-la-Gaillarde
  - CH privé St. Martin, Caen
  - CHI de Castres, Castres
  - Polyclinique Sévigné, Cesson-Sévigné
  - Hôpital Fontenoy, Chartres
  - CH Cherbourg, Cherbourg
  - CH DAX, Dax
  - CHG de Dinan, Dinan
  - Clinique Notre Dame, Draguignan
  - Polyclinique Louis Pasteur, Essey-lès-Nancy
  - CHG Saint Louis - SIH Eure Seine, Évreux
  - CHU Albert Michalon, Grenoble
  - Casamance, La Ciotat
  - CH de La Roche sur Yon, La Roche-sur-Yon
  - CH de Laval, Laval
  - Polyclinique du Bois, Lille
  - Hôpital Nord, Marseille
  - CH Emile Muller, Mulhouse
  - Nouvelles Cliniques Nantaises, Nantes
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - CH Nevers, Nevers
  - CHU Nîmes, Nîmes
  - Clinique A. Brillard, Nogent-sur-Marne
  - CHR la Source, Orléans
  - CHG de Pau, Pau
  - CH Maréchal Joffre, Perpignan
  - Clinique St Hilaire, Rouen
  - CHP de la Loire, Saint-Etienne
  - Clinique Belledone, Saint-Martin-d'Hères
  - Clinique de L'Ormeau, Tarbes
  - Clinique Pasteur, Toulouse
  - Hôpital de Brabois, Vandœuvre-lès-Nancy
- CHU de Point à pitre, Pointe-à-Pitre, Guadeloupe